CLINICAL TRIAL: NCT03470532
Title: Comparing the Effect of 4% Articaine and 2% Mepivacaine Without Palatal Injection in Pain Assessment During Maxillary Teeth Extraction- A Randomized Clinical Trial
Brief Title: Comparing Articaine and Mepivacaine Without Palatal Injection in Pain Assessment During Maxillary Teeth Extraction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Melaka Manipal Medical College (Other)
Responsible Party: Principal Investigator, Abdul Kalam Azad, Assistant Professor, Dept Of Oral and Maxillofacial Surgery, Melaka Manipal Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MMMC/FOD/AR/B5/E C-2017(24)
Record Dates: First submitted 2018-03-09; First posted 2018-03-20 (Actual); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Carticaine; Epinephrine; Mepivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (Experimental): buccal infiltration of 4% Articaine with epinephrine
  Interventions: Drug: buccal infiltration of 4% Articaine with Epinephrine
- Group B (Active Comparator): buccal infiltration of 2% Mepivacaine with epinephrine
  Interventions: Drug: buccal infiltration of 2% Mepivacaine with Epinephrine

INTERVENTIONS:
Drug: buccal infiltration of 4% Articaine with Epinephrine — Articaine Hydrochloride 4 % / Epinephrine 1:200,000 1.8 ML Cartridge
  Other Names: Septocaine 4%
  Arms: Group A
Drug: buccal infiltration of 2% Mepivacaine with Epinephrine — Mepivacaine Hydrochloride 2% Epinephrine 1:200,000 2.2 Ml Cartridge
  Other Names: Scandonest 2%
  Arms: Group B

SUMMARY:
This study compares the the efficacy of buccal infiltration of 4% Articaine and 2% Mepivacaine without any palatal injection during extraction of maxillary teeth. One group of patient receives buccal infiltration of Articaine and another group receives buccal infiltration of Mepivacaine.

DETAILED DESCRIPTION:
Dense local anesthesia is required to reduce pain during extraction of tooth. Administration of local anesthesia to the palatal mucosa is proved to be the most painful due to its firm adherence to the underlying periosteum and also it's abundant nerve supply. Articaine has greater lipid solubility and high bone penetration property. Mepivacaine is proven to be the safest local anaesthetic agent. Avoidance of a palatal injection during extraction will benefit the patient by reducing pain and anxiety to a greater extent.

So this study compares the bone penetration property between Articaine and Mepivacaine by assessing the pain in the palatal mucosa while extracting the tooth using only buccal infiltration.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and above
* Patients requiring extraction of maxillary teeth which are grossly decayed, grade I mobile, root stumps or indicated for therapeutic extractions.
* Healthy patients ( ASA I ) or patients with mild systemic disease with no functional limitations (ASA II).
* Patients who are not allergic to the drugs used in the study

Exclusion Criteria:

* Patients with periapical infections.
* Patients who are on concurrent treatment with NSAIDs and corticosteroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-02-25 (Actual); Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Measurement of pain intensity | 10 minutes after the administration of the drug
  pain intensity in the palatal mucosa is measured using Visual Analogue Scale during instrumentation to check objective symptoms of numbness. The pain is marked from 0-100 mm in a 100 mm visual analogue scale ( 0= no pain, 100= extremely severe pain).
Measurement of pain intensity | through the extraction procedure
  pain intensity in the palatal mucosa is measured using Visual Analogue Scale during flap elevation procedure . The pain is marked from 0-100 mm in a 100 mm visual analogue scale ( 0= no pain, 100= extremely severe pain).
Measurement of pain intensity | Through the extraction procedure
  pain intensity is measured using Visual Analogue Scale during extraction of tooth. The pain is marked from 0-100 mm in a 100 mm visul analogue scale ( 0= no pain, 100= extremely severe pain).

SECONDARY OUTCOMES:
Response rate | Through the extraction procedure
  the total number of patients with pain score more than 40 mm in visual Analogue Scale resulting in a palatal injection.

CONTACTS AND LOCATIONS:
Overall Officials: Abdul k Azad, MDS, Principal Investigator — Melaka Manipal Medical College,Faculty of Dentistry, Manipal Academy of Higher Education
Locations (1):
- Melaka Manipal Medical College, Malacca, Malaysia